CLINICAL TRIAL: NCT06143943
Title: Anterior Segment Anatomic Parameters Based on the Scleral Spur and Cornea for Risk Profiling of Primary Angle-closure Glaucoma
Brief Title: Anterior Segment Anatomic Parameters for Risk Profiling of Primary Angle-closure Glaucoma
Status: Completed | Type: Observational
Sponsor: Min Ke (Other)
Responsible Party: Sponsor-Investigator, Min Ke, Professor of Treatment, Zhongnan Hospital
Organization: Zhongnan Hospital (Other)
Other Study IDs: 20231116
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Glaucoma, Angle-Closure
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- primary angle-closure glaucoma
- narrow angle

SUMMARY:
The goal of this observational study is to examine the anterior segment anatomical parameters associated with the scleral spur and cornea for risk profiling of primary angle-closure glaucoma (PACG). The main question it aims to answer is:

• Are there new anatomical parameters of the anterior segment of the eye that can be used early for risk profiling for PACG? Researchers will compare PACG and narrow angle groups to see if there are some anatomical parameters that can distinguish the two.

DETAILED DESCRIPTION:
We aimed to examine the anterior segment anatomical parameters associated with the scleral spur and cornea for risk profiling of primary angle-closure glaucoma (PACG).

This retrospective study included 84 patients with PACG and 84 patients with narrow angles (NA). We collected parametric measurements obtained using anterior-segment optical coherence tomography and IOLMaster 700. Univariate and multivariate logistic regression models were used to compare the ocular parameters between the NA and PACG groups as well as to identify risk factors for PACG. The predictive performance of each parameter was evaluated using the area under the receiver operating characteristic curve (AUROC) analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Primary angle-closure glaucoma （PACG) was defined as an occlusion angle with peripheral anterior synechiae and intraocular pressure (IOP) > 21 mmHg or associated with glaucomatous optic neuropathy. The following conditions were identified as possible glaucomatous optic neuropathies, including a vertical cup-to-disc ratio ≥ 0.6, vertical cup-to-disc ratio asymmetry ≥ 0.2, optic disc haemorrhage, and visible retinal nerve fibre layer defect.
2. Participants with narrow angle (NA) were selected from among patients with cataracts. NA was defined as a trabecular-iris angle (TIA) < 15° on anterior segment optical coherence tomography, with the exclusion of glaucomatous optic neuropathy or visual field loss.

Exclusion Criteria:

(1) severe systemic disease, (2) secondary angle-closure glaucoma, (3) other ocular diseases, (4) history of intraocular surgery, and (5) unclear examination images.

Ages: 30 Years to 92 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PACG and anterior chamber angle stenosis were enrolled in this study and excluded from other diseases affecting the structure of the anterior segment of the eye, as well as a history of intraocular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Trabecular scleral-spur angle | 2022-11-22 to 2022-12.31
  The angle between the line of the corneal endothelium 750 μm from the scleral spur to the scleral spur and the bilateral line of the scleral spur

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No